CLINICAL TRIAL: NCT04305808
Title: Characterization of Vaginal, Urinary and Fecal Microbiomes in Women with Recurrent Urinary Tract Infections
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, MD, Hadassah Medical Organization
Other Study IDs: 0014-20-HMO
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Urinary Tract Infections; Menopause
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal, urine and fecal samples for microbiome molecular analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recurrent Urinary tract infection: Menopausal women, with two or more documented, culture-positive infections in the last six months or ≥3 infections in the last year
- Healthy controls: Menopausal women, without prior history of UTIs or other urologic abnormalities.

SUMMARY:
The objectives are to evaluate whether variations in vaginal and/or urinary and/or fecal microbiome predispose postmenopausal women to recurrent cystitis. This will be explored using comparison of microbiome profiles between those with recurrent UTI compared to age-matched women without recurrent UTI.

DETAILED DESCRIPTION:
Patients and age-matched control subjects will be recruited from the Urogynecology clinic in Hadassah Mt Scopus and the gynecology clinic, respectively.

After assessment of inclusion and exclusion criteria and patient's consent to participate, a history intake (detailing demographics, medical history, risk factors for rUTI etc.) and gynecological examination will be conducted as part of the usual assessment in the clinic.

Vaginal, urine and fecal samples for microbiome molecular analysis will be collected during clinic visits, given at least one month without antibiotics before samples collection, using agreed protocols and will be kept for future evaluation. Urine will be collected for urinalysis and for a urine culture.

In addition, urine cultures, as well as vaginal, urine and fecal samples for molecular analysis will be collected during an acute UTI episode from the same patients.

Healthy patients (the control group) will be examined only once.

ELIGIBILITY:
Patients' inclusion criteria:

* Menopausal status
* Two or more documented, culture-positive infections in the last six months or ≥3 infections in the last year Patients' exclusion criteria
* Neurogenic bladder condition
* Known immunodeficiencies
* Usage of antibiotics or probiotics within the previous month
* Known renal calculi or anatomic malformations

Control subjects- Inclusion criteria:

* Menopausal status
* Sterile urine cultures, normal urinalysis, and negative sexually-transmitted PCR urine assay

Control subjects- Exclusion criteria:

- A prior history of UTIs or other urologic abnormalities.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Menopausal women, with recurrent UTI and age-matched menopausal women without recurrent UTI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of the microbiome using molecular methods. | 1 year
  Comparison of microbiome profiles between those with rUTI compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No